CLINICAL TRIAL: NCT01586026
Title: A Retrospective Study to Extend the Maximum Maintenance Flushing Interval for Ports With Distally Valved Catheters
Brief Title: Study to Extend the Maximum Maintenance Flushing Interval for Ports With Distally Valved Catheters
Acronym: DISTAL
Status: Terminated | Type: Observational
Why Stopped: Insufficient number of adverse events
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Other Study IDs: BAS-11-001
Record Dates: First submitted 2012-04-25; First posted 2012-04-26 (Estimated); Results first posted 2016-08-23 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-07

CONDITIONS: Cancer
Keywords: Ports; Catheters; Distal Valved Catheters; Maintenance Flush; subjects; routine maintenance flushes
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group A: Maintenance flushes at days 1-28
- Group B: Maintenance flushes at days 29-56
- Group C: Maintenance flushes at days 57+

SUMMARY:
This study is to compare the rate of adverse events in subjects with maintenance flushes greater than 28 days.

DETAILED DESCRIPTION:
This study is a retrospective, multi-center data collection study to support extending the maximum recommended maintenance flushing intervals in subjects who have Bard totally implanted ports with distally-valved catheters.

This study is intended to provide clinical evidence in support of extending the maximum recommended maintenance flushing interval to a time point of potentially >28 days for Bard ports with distally-valved catheters.

Reduction in the number of maintenance flushes could help alleviate the inconvenience, reduce the time and expense, and minimize the invasive nature of the maintenance flushing procedure for patients and medical institutions. Subjects will be eligible for analysis of the primary endpoint after the first successful maintenance flush of the port until (a) the first adverse event or (b) abandonment of the port.

A financial analysis will be performed on an institutional basis to determine the approximate mean cost of flushing. These costs will be extrapolated into an approximate per-patient cost for the different flushing period durations. No financial information will be collected from subject medical records. All required information will be extrapolated from site staff.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 21 years
* Subject has an implanted Bard port with a distally-valved catheter
* Subject has maintenance port flushes with heparin/heparinized saline or normal saline
* Subject is post infusional cancer therapy (solid tumor or hematologic)
* Subject has signed a HIPAA Authorization to use and disclose PHI

Exclusion Criteria:

* Subject is having port maintenance flushes/locks with citrate.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects with an implanted Bard port with a distally valved catheter
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael McNamara, MD, Principal Investigator — Alegent Health
Locations (5):
- United States (5):
  - Quincy Medical Group, Quincy, Illinois
  - Willis Knighton Cancer Center, Shreveport, Louisiana
  - St. Luke's Hospital, Chesterfield, Missouri
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Alegent Research Center, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No
Study was terminated due to limited number of adverse events recorded.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 350 | 414 | 271
Completed | 350 | 414 | 271
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Post-infusional chemotherapy subjects that had Bard implanted ports with distally valved catheters.
Groups:
- Combined Demographics: Demographics of 171 subjects that contributed to final data analysis
Arm/Group | Combined Demographics
Number analyzed (Participants) | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111
  Male | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 160
  More than one race | 0
  Unknown or Not Reported | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 168
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 171
Cancer Type [Number; unit: participants]
  Solid tumor | 142
  Hematologic | 29
Port Access Vein [Number; unit: participants]
  Jugular | 65
  Subclavian | 102
  Unknown | 4
Port Configuration [Number; unit: participants]
  Single Lumen | 132
  Dual Lumen | 1
  Unknown | 38
Catheter Configuration [Number; unit: participants] — #Fr. (French units) refers to the functional lumen/relative size of the catheter's diameter with smaller numbers indicating smaller diameters. Each increment of French sizing equals 0.33 mm.
  participants
    7Fr. | 0
    8Fr. | 11
    9.5Fr. | 0
    Unknown | 160

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Adverse Events in Group A (1-28 Day Flushing Interval) Versus Extended Accession Intervals in Group B (29-56 Day Flushing Interval), and Group C (57+ Days).
Description: Subjects' maintenance flush intervals were collected by calculating the number of days since a previous flush. A total of 1,035 maintenance flush intervals were recorded at all sites. The numbers of flushing intervals available for analysis are 1,035 representing 49,696 patient days were recorded in 171 subjects.
Time Frame: 100 days
Measure: Number; unit: adverse events
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 350 | 414 | 271
adverse events | 0 | 1 | 2

ADVERSE EVENTS:
Time Frame: During retrospective review of subject records all defined adverse events were recorded from January 1, 2008 to date of chart review.
Description: Adverse events were assessed separately for each flushing interval, and not for each participant
Arm/Group | Group A | Group B | Group C
Serious Adverse Events (participants affected / at risk) | 0/350 | 0/414 | 0/271
Other Adverse Events (participants affected / at risk) | 0/350 | 1/414 | 2/271
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=350) | Group B (N=414) | Group C (N=271)
Port/Catheter Malfunction (Injury, poisoning and procedural complications) | 0 | 1 | 1 — Port would not allow for infusion of withdrawal of blood. CathFlo was administered and port functioned properly.
Fractured Catheter (General disorders) | 0 | 0 | 1 — The subject had pain radiating down the inside of the right arm during flushing. Flushing stopped and chest x-ray revealed a fractured catheter.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No